CLINICAL TRIAL: NCT01612650
Title: Assessment of Substitution of Focused Cliches and Ultrasound for Tomosynthesis
Acronym: TOMOSEIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TOMOSEIN-1104; 2011-002051-34 (Other: IDRCB number (ANSM))
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer; 2D Mammography; 3D Mammography
Keywords: breast cancer; surveillance; diagnosis; 2D mammography; 3D mammography
MeSH Terms: conditions — Breast Neoplasms; Disease | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- breast cancer histologically proven (Active Comparator): Patient with breast cancer histologically proven, addressed to Oscar Lambret Center for treatment
  Interventions: Device: tomosynthesis; Device: 2D mammography
- surveillance of a treated breast cancer (Active Comparator): surveillance of patient already treated for breast cancer must have annual mammography
  Interventions: Device: tomosynthesis; Device: 2D mammography
- diagnosis of a detected anomaly (Active Comparator): patient addressed for diagnosis of a detected anomaly
  Interventions: Device: tomosynthesis; Device: 2D mammography

INTERVENTIONS:
Device: tomosynthesis — 2 incidences 3D numeric mammography
Device: 2D mammography — 2 incidences 2D analogic mammography

SUMMARY:
This study aims to assess if using tomosynthesis for breast cancer surveillance will allow a significant decrease of ultrasound cliches (and radiation exposure)

ELIGIBILITY:
Inclusion Criteria:

* woman with breast cancer histologically proven (group 1), on surveillance of a treated breast cancer (group 2) or diagnosis of an detected anomaly
* age ≥ 40 years (group 1, group 2); age ≥ 50 years (group 3)
* breast size suitable for detector size
* possible prior mastectomy
* security social covered
* signed informed consent

Exclusion Criteria:

* breast implant
* high genetic risk (mutation)
* under justice measures
* breast feeding or pregnant woman

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1069 (Actual)
Dates: Start 2012-02-24 (Actual); Primary Completion 2017-03-16 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
determine the benefit of tomosynthesis for diagnosis | 30 months
  number of avoided focused cliches and ultrasound, after tomosynthesis analysis

SECONDARY OUTCOMES:
determine best incidence of realization | 30 months
  face, medial side or oblique
measurement of breast irradiation | 30 months
  comparison of tomosynthesis irradiation and focused cliches irradiation
evaluate non focused ultrasound residual place for 2 - 3 - 4 density breast | 30 months
number of additional cancer detected by tomosynthesis | 30 months
  number of breast cancer detected through tomosynthesis

CONTACTS AND LOCATIONS:
Overall Officials: Sophie TAIEB, MD, Principal Investigator — Oscar Lambret Center
Locations (4):
- France (4):
  - Oscar Lambret Center, Lille
  - Centre Hospitalier - Pavillon Paul Gelé, Roubaix
  - Centre Hospitalier, Valenciennes
  - Clinique des Dentellières, Valenciennes

IPD SHARING:
Plan to Share IPD: No